CLINICAL TRIAL: NCT06237803
Title: EMN Prospective Sample Collection Project
Brief Title: European Myeloma Network (EMN) Sample Project
Acronym: EMN36
Status: Recruiting | Type: Observational
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: EMN36
Record Dates: First submitted 2024-01-15; First posted 2024-02-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma; Smoldering Multiple Myeloma; Plasma Cell Leukemia; Extramedullary Myeloma; MGUS
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma; Leukemia, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * bone marrow aspirate, bone marrow biopsy, extramedullary disease (EMD) biopsy, peripheral blood and serum at baseline;
  * bone marrow aspirate, bone marrow biopsy, peripheral blood and serum pre-maintenance in TE patients or after 1 year of therapy in non transplant eligible patients;
  * bone marrow aspirate, bone marrow biopsy, peripheral blood and serum during maintenance therapy and only if performed as standard of care (SOC);
  * bone marrow aspirate, bone marrow biopsy, EMD biopsy peripheral blood and serum at 1st and later progressive disease (PD).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with MGUS, SMM, MM, PCL: Subjects with Monoclonal Gammopathy of Undetermined Significance (MGUS), smouldering Multiple Myeloma (SMM), Multiple Myeloma (MM), Plasma Cell Leukemia (PCL)
  Timepoints and samples to be collected are the following:
  * bone marrow aspirate, bone marrow biopsy, EMD biopsy, peripheral blood and serum at baseline;
  * bone marrow aspirate, bone marrow biopsy, peripheral blood and serum pre-maintenance in TE patients or after 1 year of therapy in Non-Transplant-Eligible (NTE) patients;
  * bone marrow aspirate, bone marrow biopsy, peripheral blood and serum during maintenance therapy and only if performed as SOC;
  * bone marrow aspirate, bone marrow biopsy, EMD biopsy peripheral blood and serum at 1st and later PD.
  Interventions: Other: storage of biological samples

INTERVENTIONS:
Other: storage of biological samples — collect and store biological samples

SUMMARY:
This is an observational, non-interventional, multicenter study for the prospective collection, storage and analysis of patients' biological samples.

This study establishes a common international infrastructure useful to collect standard clinical variables at baseline and during treatment and to uniformly collect and store biological samples

ELIGIBILITY:
Inclusion Criteria:

* Subjects with MGUS, smouldering Multiple Myeloma (SMM) , MM (Multiple Myeloma) (+/- EMD), plasma cell leukemia (PCL) (+/- EMD)
* Subjects are ≥ 18 years old.
* Subjects have provided written informed consent in accordance with federal, local, and institutional guidelines prior to initiation of any project-specific activities or procedures.

  1. Subjects do not have kind of condition that, in the opinion of the Investigators, may compromise the ability of the subjects to give written informed consent and
  2. subjects are, in the investigator's opinion, willing and able to comply with the protocol requirements.

Exclusion Criteria:

* Previous treatment with anti-myeloma therapy (excluding one course of therapy in patients in which urgent therapy is deemed necessary according to physician's discretion, e.g. myeloma-related complications resistant to supportive care).
* Subjects have had prior unforeseen (serious) adverse reactions to blood donation including, but not limited to fainting, angina, severe bruising, allergic reactions, or any other adverse events.
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in hospitals in countries that participate in European Myeloma Network (EMN) trials; these patients may be included in upfront trials or in maintenance or relapse trials later during their disease.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2037-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Biobank | up to 30 years
  Collect biological samples for research studies related to improving medicine and care to the patient

CONTACTS AND LOCATIONS:
Locations (41):
- Alfred Hospital, Melbourne, Australia
- Austria (2):
  - KUK Linz, Linz
  - Medical University Vienna, Vienna
- Department of Haematology UZ Leuven Gasthuisberg, Leuven, Belgium
- Czechia (7):
  - Nemocnice Havířov, Havířov
  - Nemocnice Nový Jičín, Nový Jičín
  - Fakultní nemocnice, Olomouc
  - Slezská nemocnice, Opava
  - Fakutni nemocnice Ostrava, Ostrava
  - Nemocnice Pelhrimov, Pelhřimov
  - Všeobecná Fakultní nemocnice v Praz, Prague
- Greece (2):
  - Regional General Hospital Alexandra Dept of Clinical Therapeutics, Athens
  - Theagenion Cancer Hospital, Thessaloniki
- Beaumont Hospital, Dublin, Hematology Department, Galway, Ireland
- Italy (20):
  - A.O. 'SS. Antonio e Biagio', Alessandria
  - AOU Ospedali Riuniti di Ancona, Ancona
  - Bari-A.O.U. Consorziale Policlinico - Medicina Interna, Bari
  - Policlinico S Orsola Malpighi, Bologna
  - A.O.Spedali Civili di Brescia, Brescia
  - A.S.U.R. Regione Marche, Civitanova Marche
  - A.O.U. Careggi, Florence
  - A.O.U. Policlinico S. Martino - Clinica Ematologica, Genova
  - A.O.U. Policlinico S. Martino - Ematologia, Genova
  - A.O. 'Cardinale G.Panico', Lecce
  - A.O. di Rilievo Nazionale A. Cardarelli, Napoli
  - A.O.U. Maggiore della Carità, Novara
  - Policlinico S. Matteo Fondazione IRCCS - Pavia, Pavia
  - A.O. San Camillo-Forlanini, Roma
  - Ospedale S. Eugenio, Roma
  - I.R.C.C.S. Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - A.O. S. Maria, Terni
  - A.O.U. Città della Salute e della Scienza di Torino - PO Molinette, Torino
  - Azienda Ospedaliera Universitaria di Udine, Udine
  - ULSS8 Berica Ospedale S.Bortolo, Vicenza
- Portugal (4):
  - CHUC, Coimbra
  - Fundação Champalimaud, Lisbon
  - Chsj - Hosp. Sao Joao, Porto
  - IPOP Porto, Porto
- Clinic of Hematology, University Clinical Center of Serbia, Belgrade, Serbia
- Switzerland (2):
  - CHUV, Lausanne
  - HOCH Health Ostschweiz Kantonsspital St.Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Undecided